CLINICAL TRIAL: NCT06155201
Title: To Develop Intelligent Warning, Diagnosis and Intervention Systems for Children and Adolescents With Mental Disorders and Developmental Behavioral Disorders
Brief Title: Development and Application of Intelligent Diagnosis and Treatment Norms for Children and Adolescents With Mental Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Li (Other)
Collaborators: Southwest University, China (Unknown); Sichuan University ，China (Unknown); First Affiliated Hospital of Chongqing Medical University (Other); Dachuan District People's Hospital，China (Unknown); Chongqing Beiminglian Digital Technology Co. LTD，China (Unknown)
Responsible Party: Sponsor-Investigator, Chen Li, Associate Professor, Director, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IDTSDA
Record Dates: First submitted 2023-11-17; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Depressive Disorder; AD; ASD; ADHD
Keywords: intelligence diagnosis and treatment system; Depressive Disorder; AD; ASD; ADHD
MeSH Terms: conditions — Depressive Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Observation

STUDY DESIGN:
Intervention Model Description: Collect blood samples from more than 5,000 patients with depression, more than 5,000 patients with anxiety disorders, more than1000 patients with autism spectrum disorder, and more than1000 patients with attention deficit hyperactivity disorder, and complete different intervention for a total of more than 12,000 patients. Based on the CCBT theory Moca system and systematic aerobic exercise system and other projects, personalized functional training intervention for children can be achieved. Use wearable diagnostic and treatment equipment, such as brain imaging, brain functional imaging, and neuromodulation technology to assist diagnosis and treatment; use structured psychological behavioral therapy and artificial intelligence technology to improve management.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- depression disorder (Experimental): The depressive disorder group must complete four years of follow-up and intervention. Collect blood samples from more than 5,000 patients with depressive disorders.
  Interventions: Behavioral: functional training; Other: Observation
- anxiety disorder (Experimental): The anxiety disorder group must complete four years of follow-up and intervention. Collect blood samples from more than 5,000 patients with depressive disorders.
  Interventions: Behavioral: functional training; Other: Observation
- autism spectrum disorder (Experimental): The autism spectrum disorder group must complete four years of follow-up and intervention. Collect blood samples from more than 1,000 patients with depressive disorders.
  Interventions: Behavioral: functional training; Other: Observation
- attention deficit hyperactivity disorder (Experimental): The attention deficit hyperactivity disorder group must complete four years of follow-up and intervention. Collect blood samples from more than 1,000 patients with depressive disorders.
  Interventions: Behavioral: functional training; Other: Observation

INTERVENTIONS:
Behavioral: functional training — Based on individual differences, children are provided with structural psychological behavioral therapy, including the implementation of aerobic exercise and executive skills training based on motivational quotient theory. Use brain imaging, brain functional imaging and neuromodulation technology to improve children's symptoms.
Other: Observation — Children with depressive disorders, anxiety disorders, autism spectrum disorders, and attention deficit hyperactivity disorder were recruited at presentation. Differential interventions and assessments were conducted during the study.

SUMMARY:
The prevalence of mental disorders and developmental behavioral disorders (such as depressive disorders,anxiety disorders, autism spectrum disorders,attention deficit disorder,ect.)among children and adolescents in China is increasing,leading to difficulty in early identification of children and poor diagnosis and treatment effects,which brings significant financial burden to the families and the country.We will carry out a multi-center epidemiological survey on common mental disorders above among children and adolescents in Sichuan-Chongqing region and clarify the prevalence,geographical distribution and demographic characteristics.A total of more than 12,000 children and adolescents under 18 years old with a diagnosis of depression/anxiety disorders/ASD/ADHD based on DSM-5 criteria is included to build a research platform and database,so that we will formulate intelligence diagnosis and treatment standards.This study will establish the "Children and Adolescents Mental and Developmental Disabilities Innovation Alliance" in Sichuan and Chongqing areas and finally build intelligent early warning,diagnosis and intervention systems for disease in hope that technology transformation to be promoted and applied.

DETAILED DESCRIPTION:
1. Procedures. From January 2023 to December 2023,obtain the number of primary school students in the nine economic zones of Sichuan and Chongqing, and calculate the proportion of primary school students in each region. Randomly select 2-3 classes from each school's grade (determined based on the proportion of primary school students in each functional region and class size), and use class clusters as the research object. Establish the "Children and Adolescents Mental and Developmental Disabilities Innovation Alliance" in Sichuan and Chongqing areas.From January 2023 to December 2025,finish collecting the required sample size for four types of mental and psychological disorders. Bring into children and adolescents who meet the standards and build the epidemiological database. Develop and continuously improve different intervention plans for Moca and systematic aerobic exercise training in patients with DD, AD, ASD, and ADHD, and apply neuroregulatory techniques to evaluate and treat the aforementioned diseases.During 2025,build intelligent early warning,diagnosis and intervention systems for disease.Finally promote the application of databases and intelligent diagnosis and treatment systems in multiple institutions in more than 10 districts and counties in Sichuan-Chongqing region,with no less than 500 users per unit.
2. Demographic questionnaire and clinical data. The demographic questionnaire is completed by the child's primary caregiver, detailing child's name, gender, date of birth, height, weight, blood pressure, heart rate. Clinical data will be ascertained from the medical records, including information about DSM-5 diagnosis, disease classification, current treatment, and comorbid conditions.
3. Sample size.This study is an interventional trial. The total number of samples in the database reached>12000. Among them, the total number of depressive disorders reached>5000, the total number of anxiety disorders reached>5000, the total number of autism spectrum disorders reached>1000, and the total number of attention deficit hyperactivity disorder reached>1000. Children with depressive disorders, anxiety disorders, autism spectrum disorders, and attention deficit hyperactivity disorder are required to complete four years of follow-up and intervention. Blood samples will also need to be collected from each child included in the database. Adopt a set of wearable diagnosis and treatment equipment for common mental, psychological and developmental behavioral disorders in children and adolescents, and establish an auxiliary diagnosis and treatment system through brain imaging, brain function imaging, and neuromodulation technology. At the same time, differentiated intervention is carried out in aerobic exercise, quotient theory, and executive skills training, supplemented by the CCBT theory Moca system, structured psychotherapy and artificial intelligence technology, and combined with the auxiliary diagnosis and treatment system to build an intelligent early warning, diagnosis and intervention system.
4. Statistical analysis.All the data are analyzed using SPSS 25.0 or R language,which enters by a dedicated person,and checks by three people to ensure accurate data entry.Statistical analysis is completed under the guidance of professional statistical analysts from the Epidemiology Research Office of the project leader's unit.
5. Ethical matters and data protection. Before epidemiological survey,children and guardians participating in the study signed a consent form and schools signed a disclaimer.During the study,medical ethics laws and regulations were strictly observed,and psychiatrists,psychologists and pediatricians participated in the entire process to provide health protection for children.And they protect the privacy of subjects and do not disclose subjects' information.

ELIGIBILITY:
Inclusion Criteria:

* Depression patients:(1)Diagnose of depression according to DSM-5;Having the ability to act independently;Clear awareness;Able to communicate normally;Consent to the study ; (2)Under 18 years old;
* Anxiety patients: (1)Diagnose of anxiety according to DSM-5;Having the ability to act independently;Clear awareness;Able to communicate normally;Consent to the study ; (2)Under 18 years old;
* ASD patients:(1) Diagnose of ASD according to DSM-5;Do not have other neurological developmental disorders; (2)Under 18 years old;
* ADHD patients: (1) Diagnose of ADHD according to DSM-5;Do not have other neurological developmental disorders; (2)Aged 4-18 years old;

Exclusion Criteria:

* suffering other mental illnesses and neurological disorders now or in the past
* suffering severe physical illnesses now or in the past
* substance or drug abuse now or in the past

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the Vanderbilt Assessment Scale | 2 years
  The use of the Vanderbilt Assessment Scale scores in follow-up visits every three months reflects the ADHD symptomatology of children at different follow-up milestones. The total score of the Vanderbilt Assessment Scale can range from 0 to 54. A higher score indicates a greater likelihood of ADHD symptoms or difficulties with attention and behavior.
Changes in the Social Responsive Scale(SRS). | 3 years
  Children are followed up every 3 months, and at each follow-up point, the SRS is used to assess a child's level of social sensitivity and interpersonal skills. The SRS score ranges from 0 to 68, where 0 to 15 is considered low risk, 16 to 30 is considered medium risk, and 31 to 68 is considered high risk.
Changes in the Autism Behavior Scale(ABC). | 3 years
  Conducting follow-up assessments every 3 months using the Autism Behavior Scale (ABC) scores reflect five dimensions, including sensation, communication, body movement, language and self-care. The total score ranges from 0 to 158. Higher scores may indicate that the child has more severe symptoms of developmental disorders such as autism.
Changes in Questionnaire-Children with Difficulties（QCD） | 3 years
  Follow-up assessments every 3 months, using the Questionnaire-Children with Difficulties (QCD) scores, reflect children's psychological issues and behavioral difficulties. The scoring range of the QCD questionnaire may vary depending on the specific version or rating system. For example, certain rating systems may categorize scores into levels of severity such as mild, moderate, or severe difficulties. Higher scores may indicate higher levels of psychological difficulties or disorders. Conversely, lower scores may suggest fewer problems or mild manifestations.
Changes in the Child Anxiety Related Emotional Disorders Scale（SCARED）. | 3 years
  Conducting follow-up assessments every 3 months using the Child Anxiety Related Emotional Disorders Scale（SCARED）scores reflect children's anxiety symptoms mainly from five dimensions: somatization/panic, generalized anxiety, dissociative anxiety, social phobia, and school phobia of children at different follow-up points. Score 0-3 ("not at all" is 0, "sometimes" is 1, and "very often" is 2). Scores greater than or equal to 23 indicate the possibility of anxiety.The higher the score, the higher the level of anxiety.
Change in the Parenting Stress Index(PSI). | 3 years
  Conducting follow-up assessments every 3 months using the Parenting Stress Index (PSI) ,which is a popular brief assessment of parenting stress. The higher score indicates more anxious the parents are.
Change in the Children's Sleep Habits Questionnaire (CSHQ). | 3 years
  Conducting follow-up assessments every 3 months using the Children's Sleep Habits Questionnaire (CSHQ) score reflects key sleep domains that encompass the major medical and behavioral sleep disorders. It's a useful sleep screening instrument to identify both behaviorally based and medically-based sleep problems in school-aged children, which could get the children's sleep time, total score of sleep quality and scores of eight dimensions. A total score higher than 54 points indicates poor sleep quality.
Change in the Epidemiological Studies Depression Scale for Children (CES-DC) . | 3 years
  CES-DC is specially designed to evaluate the frequency of current depressive symptoms in children. It focuses on depressive affect or mood, reflecting the depressive mood, guilt and worthlessness, helplessness and hopelessness, and psychomotor retardation of the depressive state. , loss of appetite, sleep disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, doctor, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Growth,Development and Mental Health of Children and Adolescents Center, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study.